CLINICAL TRIAL: NCT01920126
Title: The Effect of Sodium Bicarbonate on Postoperative Renal Function in Infective Endocarditis Patients Undergoing Open Heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2013-0376
Record Dates: First submitted 2013-07-31; First posted 2013-08-09 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Acute Kidney Injury
Keywords: sodium bicarbonate, renal function, infective endocarditis, open heart surgery
MeSH Terms: conditions — Acute Kidney Injury; Endocarditis | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium bicarbonate group (Experimental): Sodium bicarbonate group
  Interventions: Drug: sodium bicarbonate
- Saline group (Placebo Comparator): Saline group
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: sodium bicarbonate — 0.5 mmol/kg for 1 hr, and then 0.15 mmol/kg/h for 23 hrs The infusion of study drug is started after anesthesia induction and continued until 24 hours after surgery
  Arms: Sodium bicarbonate group
Drug: Saline
  Arms: Saline group

SUMMARY:
The purpose of study is to test whether perioperative sodium bicarbonate infusion can prevent acute kidney injury following open heart surgery in infective endocarditis patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients over the age of 20 scheduled for open heart surgery for infective endocarditis

Exclusion Criteria:

* end stage renal disease (serum creatinine concentration > 300 μmol/L)
* on dialysis
* chronic moderate to high dose corticosteroid therapy (> 10 mg/day prednisolon or equivalent)
* preoperative severe hypernatremia (Na+ > 150 mmol/L), alkalemia (PH > 7.50), or pulmonary edema
* neurocognitive dysfunction

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2016-08-23 (Actual); Study Completion 2016-08-23 (Actual)

PRIMARY OUTCOMES:
Comparison of the the peak creatinine level during the postoperative 48h by more than 0.3 mg/dL between two groups. | postoperative 48 hours
  We would investigate if the peak creatinine level during the postoperative 48h would differ by more than 0.3 mg/dL between two groups. The primary outcome was decided based on the AKIN criteria which defines acute kidney injury if serum creatinine increases more than 0.3 mg/dL during the postoperative 48 h.
  ; increase in serum creatinine of 0.3 mg/dL or >50 percent developing over <48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Cho JS, Soh S, Shim JK, Kang S, Choi H, Kwak YL. Effect of perioperative sodium bicarbonate administration on renal function following cardiac surgery for infective endocarditis: a randomized, placebo-controlled trial. Crit Care. 2017 Jan 5;21(1):3. doi: 10.1186/s13054-016-1591-z. PMID 28057030